CLINICAL TRIAL: NCT03945292
Title: A Placebo-Controlled, Multi-dose, Phase 2 Study to Determine the Safety, Tolerability and Pharmacodynamic Effect of Fazirsiran (TAK-999, ARO-AAT) in Patients With Alpha-1 Antitrypsin Deficiency (AATD) [SEQUOIA]
Brief Title: Safety, Tolerability and Pharmacodynamic Effect of Fazirsiran (TAK-999, ARO-AAT)
Acronym: SEQUOIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAAT2001; 2018-003385-14 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Fazirsiran 25 mg DB/200 mg OL (Experimental): Double-blind (DB) Period: Participants with no fibrosis: Administered on Day 1 and Week 4. Participants with fibrosis: Administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
  Open-label (OL) Period: Participants with fibrosis at Screening who received double-blind (DB) fazirsiran 25 mg and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
  Interventions: Drug: Fazisiran Injection
- Fazirsiran 100 mg DB/200 mg OL (Experimental): DB Period: Participants with no fibrosis: Fazirsiran 100 mg administered on Day 1 and Week 4. Participants with fibrosis: Fazirsiran 100 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
  OL Period: Participants with fibrosis at Screening who received double-blind (DB) fazirsiran 100 mg and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
  Interventions: Drug: Fazisiran Injection
- Fazirsiran 200 mg DB/200 mg OL (Experimental): DB Period: Participants with no fibrosis: Fazirsiran 200 mg administered on Day 1 and Week 4.
  Participants with fibrosis: Fazirsiran 200 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
  OL Period: Participants with fibrosis at Screening who received double-blind (DB) fazirsiran 200 mg and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study
  Interventions: Drug: Fazisiran Injection
- Placebo DB / Fazirsiran 200 mg OL (Placebo Comparator): DB Period: Participants with no fibrosis: Placebo administered on Day 1 and Week 4. Participants with fibrosis: Placebo administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
  OL Period: Participants with fibrosis at Screening who received double-blind (DB) placebo and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
  Interventions: Drug: Fazisiran Injection; Other: Placebo

INTERVENTIONS:
Drug: Fazisiran Injection — solution for subcutaneous (sc) injection
  Other Names: ARO-AAT Injection; TAK-999 Injection
Other: Placebo — sterile normal saline (0.9% NaCl), calculated to match active comparator, for sc injection
  Arms: Placebo DB / Fazirsiran 200 mg OL

SUMMARY:
The purpose of AROAAT2001 (SEQUOIA) is to evaluate the safety, efficacy and tolerability of multiple doses of the investigational product, Fazirsiran Injection, administered subcutaneously to participants with alpha-1 antitrypsin deficiency (AATD).

DETAILED DESCRIPTION:
Participants will be enrolled to receive multiple subcutaneous injections of Fazirsiran Injection (also referred to as TAK-999 Injection or ARO-AAT Injection) or placebo. Eligible participants will require a pre-dose biopsy completed as part of the study within the screening window. However, any participant with a biopsy result within 1 year of screening showing no fibrosis does not require a pre-dose biopsy. Only participants who have liver fibrosis will undergo a post-dose biopsy and may continue treatment in an open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AATD
* Liver biopsy at Screening indicating liver fibrosis (score less than F4); a patient with no fibrosis may participate based on a previous biopsy conducted within one year
* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* Non-smoker for at least 1 year
* No abnormal finding of clinical relevance at Screening

Exclusion Criteria:

* Clinically significant health concerns other than AATD
* Previous diagnosis or diagnosis at Screening of definitive liver cirrhosis
* Previous lung or liver transplant due to AATD
* Regular use of alcohol within one month prior to Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study involving therapeutic intervention
* Use of illicit drugs within 1 year prior to Screening

NOTE: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (16):
  - Research Site 5, Birmingham, Alabama
  - Research Site 9, Phoenix, Arizona
  - Research Site 14, La Jolla, California
  - Research Site 17, Los Angeles, California
  - Research Site 11, Sacramento, California
  - Research Site 15, San Francisco, California
  - Research Site 13, Stanford, California
  - Research Site 2, Gainesville, Florida
  - Research Site 7, Indianapolis, Indiana
  - Research Site 3, Iowa City, Iowa
  - Research Site 10, St Louis, Missouri
  - Research Site 12, New York, New York
  - Research Site 1, Charleston, South Carolina
  - Research Site 4, Nashville, Tennessee
  - Research Site 19, Houston, Texas
  - Research Site 16, Salt Lake City, Utah
- Research Site 27, Aachen, Germany
- Research Site 22, Pavia, Italy
- Research Site 23, Leiden, Netherlands
- Research Site 24, Funchal, Portugal
- Research Site 20, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark VC, Strange C, Strnad P, Sanchez AJ, Kwo P, Pereira VM, van Hoek B, Barjaktarevic I, Corsico AG, Pons M, Goldklang M, Gray M, Kuhn B, Vargas HE, Vierling JM, Vuppalanchi R, Brantly M, Kappe N, Chang T, Schluep T, Zhou R, Hamilton J, San Martin J, Loomba R. Fazirsiran for Adults With Alpha-1 Antitrypsin Deficiency Liver Disease: A Phase 2 Placebo Controlled Trial (SEQUOIA). Gastroenterology. 2024 Oct;167(5):1008-1018.e5. doi: 10.1053/j.gastro.2024.06.028. Epub 2024 Jul 2. PMID 38964420
- [Derived] Remih K, Amzou S, Strnad P. Alpha1-antitrypsin deficiency: New therapies on the horizon. Curr Opin Pharmacol. 2021 Aug;59:149-156. doi: 10.1016/j.coph.2021.06.001. Epub 2021 Jul 10. PMID 34256305

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was performed within each dose cohort to maintain blinding due to different dose volumes in the double-blinded phase.
Groups:
- Fazirsiran 25 mg: Participants with no fibrosis: Fazirsiran 25 mg administered on Day 1 and Week 4.
  Participants with fibrosis: Fazirsiran 25 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
- Fazirsiran 100 mg: Participants with no fibrosis: Fazirsiran 100 mg administered on Day 1 and Week 4.
  Participants with fibrosis: Fazirsiran 100 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
- Fazirsiran 200 mg: Participants with no fibrosis: Fazirsiran 200 mg administered on Day 1 and Week 4.
  Participants with fibrosis: Fazirsiran 200 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
- Placebo: Participants with no fibrosis: Placebo administered on Day 1 and Week 4.
  Participants with fibrosis: Placebo administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
- Fazirsiran 25 mg DB/200 mg OL: Participants with fibrosis at Screening who received double-blind (DB) fazirsiran 25 mg and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
- Fazirsiran 100 mg DB/200 mg OL: Participants with fibrosis at Screening who received double-blind (DB) fazirsiran 100 mg and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
- Fazirsiran 200 mg DB/200 mg OL: Participants with fibrosis at Screening who received double-blind (DB) fazirsiran 200 mg and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
- Placebo DB / Fazirsiran 200 mg OL: Participants with fibrosis at Screening who received double-blind (DB) placebo and who completed the post-dose liver biopsy at Week 48 (or Week 72 or Week 96) entered the open-label phase and received fazirsiran 200 mg every 12 weeks for the duration of the study.
Period: Double-Blind (DB) Period: Weeks 0 to 48
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo | Fazirsiran 25 mg DB/200 mg OL | Fazirsiran 100 mg DB/200 mg OL | Fazirsiran 200 mg DB/200 mg OL | Placebo DB / Fazirsiran 200 mg OL
Started | 9 | 8 | 9 | 14 | 0 | 0 | 0 | 0
Completed | 8 | 8 | 7 | 14 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-Label (OL) Period: Weeks 48 to 196
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo | Fazirsiran 25 mg DB/200 mg OL | Fazirsiran 100 mg DB/200 mg OL | Fazirsiran 200 mg DB/200 mg OL | Placebo DB / Fazirsiran 200 mg OL
Started | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 9
Completed | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 9 | 14 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (15.56) | 47.9 (12.25) | 51.6 (9.44) | 57.4 (9.05) | 53.1 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 5 | 22
  Male | 4 | 2 | 3 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 9 | 7 | 9 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 8 | 9 | 14 | 40
Fibrosis Status at Screening [Count of Participants; unit: Participants]
  Fibrosis at Screening | 4 | 5 | 7 | 9 | 25
  No fibrosis at Screening | 5 | 3 | 2 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Serum Z-Alpha-1 Antitrypsin (Z-AAT) at Week 16
Time Frame: Baseline, Week 16 (+/- 2 weeks)
Population: Full Analysis Set: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change | -62.17 (4.279) | -85.39 (4.634) | -92.93 (4.341) | 4.64 (3.211)
Statistical Analysis 1: Comparison: Fazirsiran 25 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM) — From a mixed model with repeated measures, including fixed effects for treatment, week, treatment-by-week interaction, presence of metabolic syndrome, presence of NAFLD or NASH, baseline serum Z-AAT as covariate, and subject as a random effect; NAFLD=non-alcoholic fatty liver disease; NSH=non-alcoholic steatohepatitis; Difference = -66.81, 95% CI 2-sided [-77.18 to -56.45], Standard Error of Mean 5.107
Statistical Analysis 2: Comparison: Fazirsiran 100 mg vs Placebo; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference = -90.03, 95% CI 2-sided [-100.72 to -79.34], Standard Error of Mean 5.26
Statistical Analysis 3: Comparison: Fazirsiran 200 mg vs Placebo; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference = -97.57, 95% CI 2-sided [-108.21 to -86.94], Standard Error of Mean 5.24

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Double-Blind Phase
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have to have a causal relationship with this treatment. A serious adverse event (SAE) is an AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event or reaction. TEAEs/TESAEs are defined as those AEs that first occurred or worsened in severity following dose administration through end of study (EOS) or Early Termination or first dose of open-label phase fazirsiran.
Time Frame: Double Blind Phase (up to Week 48): dose administration through end of study (EOS) or Early Termination or first dose of open-label phase fazirsiran.
Population: Safety Analysis Set: All participants who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
Participants
  TEAEs | 9 | 8 | 9 | 14
  TESAEs | 0 | 0 | 2 | 3
  TEAEs Leading to Withdrawal of Study Drug | 0 | 0 | 1 | 0
  TEAEs Leading to Study Termination | 0 | 0 | 1 | 0
  TEAEs Leading to Death | 0 | 0 | 0 | 0
  TEAEs by Worst Severity: Mild | 3 | 2 | 1 | 5
  TEAEs by Worst Severity: Moderate | 6 | 6 | 6 | 6
  TEAEs by Worst Severity: Severe | 0 | 0 | 2 | 3
  TEAEs by Worst Relationship: Not Related | 7 | 4 | 5 | 6
  TEAEs by Worst Relationship: Possibly Related | 2 | 3 | 1 | 8
  TEAEs by Worst Relationship: Probably Related | 0 | 1 | 3 | 0
  TEAEs by Worst Relationship: Possibly or Probably | 2 | 4 | 4 | 8
  TEAE at Injection Site | 1 | 1 | 2 | 2

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Open-Label Phase
Description: as for outcome 2
Time Frame: From dose administration of the first dose of open-label phase fazirsiran through EOS or Early Termination (up to Week 196).
Population: Safety Analysis Set: All participants who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 5 | 9
Participants
  TEAEs | 4 | 4 | 3 | 9
  TESAEs | 1 | 1 | 1 | 1
  TEAEs Leading to Withdrawal of Study Drug | 0 | 0 | 0 | 1
  TEAEs Leading to Study Termination | 0 | 0 | 0 | 1
  TEAEs Leading to Death | 0 | 0 | 0 | 0
  TEAEs by Worst Severity: Mild | 3 | 2 | 0 | 7
  TEAEs by Worst Severity: Moderate | 0 | 1 | 3 | 1
  TEAEs by Worst Severity: Severe | 1 | 1 | 0 | 1
  TEAEs by Worst Relationship: Not Related | 2 | 0 | 3 | 7
  TEAEs by Worst Relationship: Possibly Related | 2 | 3 | 0 | 2
  TEAEs by Worst Relationship: Probably Related | 0 | 1 | 0 | 0
  TEAEs by Worst Relationship: Possibly or Probably | 2 | 4 | 0 | 2
  TEAE at Injection Site | 1 | 1 | 0 | 0

4. Secondary Outcome: Absolute Change From Baseline in Total Liver Z-AAT (Insoluble + Soluble) Protein at Post-dose Biopsy for Participants With Fibrosis
Description: Post-dose biopsy includes all post-dose biopsy collected at Week 48 or Week 72 or Week 96.
Time Frame: Baseline, Week 48 (+/- 2 weeks), or Week 72 (+/- 4 weeks), or Week 96 (+/- 4 weeks)
Population: Biopsy Analysis Set: All randomized participants who received at least one dose of study drug and had at least one central read histology biopsy result.
Measure: Mean (Standard Deviation); unit: nmol/g
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 8
nmol/g | -89.341 (94.832) | -259.892 (330.199) | -29.371 (22.867) | -4.738 (57.342)

5. Secondary Outcome: Percent Change From Baseline in Total Liver Z-AAT (Insoluble + Soluble) Protein at Post-dose Biopsy for Participants With Fibrosis
Description: Post-dose biopsy includes all post-dose biopsy collected at Week 48 or Week 72 or Week 96.
Time Frame: Baseline, Week 48 (+/- 2 weeks), or Week 72 (+/- 4 weeks), or Week 96 (+/- 4 weeks)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 8
percentage change | -86.89 (29.658) | -81.61 (29.503) | -98.16 (23.256) | 42.42 (21.133)
Statistical Analysis 1: Comparison: Fazirsiran 25 mg vs Placebo; Test type: Superiority; p = 0.0021, ANCOVA — Model based summary statistics are from an analysis of covariance (ANCOVA) model with fixed effect factors treatment group and baseline total liver Z-AAT protein as a covariate; Least Squares (LS) Mean Difference = -129.31, 95% CI 2-sided [-205.52 to -53.11], Standard Error of Mean 36.409
Statistical Analysis 2: Comparison: Fazirsiran 100 mg vs Placebo; Test type: Superiority; p = 0.0035, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -124.03, 95% CI 2-sided [-201.9 to -46.15], Standard Error of Mean 37.207
Statistical Analysis 3: Comparison: Fazirsiran 200 mg vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -140.58, 95% CI 2-sided [-205.27 to -75.89], Standard Error of Mean 30.906

6. Secondary Outcome: Absolute Change From Baseline in Liver Z-AAT Soluble Protein at Post-dose Biopsy for Participants With Fibrosis
Description: Post-dose biopsy includes all post-dose biopsy collected at Week 48 or Week 72 or Week 96.
Time Frame: Baseline, Week 48 (+/- 2 weeks), or Week 72 (+/- 4 weeks), or Week 96 (+/- 4 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nmol/g
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 8
nmol/g | -20.427 (15.042) | -109.747 (135.114) | -17.418 (4.860) | 2.300 (12.940)

7. Secondary Outcome: Percent Change From Baseline in Liver Z-AAT Soluble Protein at Post-dose Biopsy for Participants With Fibrosis
Description: Post-dose biopsy includes all post-dose biopsy collected at Week 48 or Week 72 or Week 96.
Time Frame: Baseline, Week 48 (+/- 2 weeks), or Week 72 (+/- 4 weeks), or Week 96 (+/- 4 weeks)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 8
percentage change | -75.73 (16.645) | -87.23 (17.064) | -95.71 (12.824) | 22.33 (11.890)
Statistical Analysis 1: Comparison: Fazirsiran 25 mg vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA — Model based summary statistics are from an analysis of covariance (ANCOVA) model with fixed effect factors treatment group and baseline soluble liver Z-AAT protein as a covariate; LS Mean Difference = -98.07, 95% CI 2-sided [-140.53 to -55.6], Standard Error of Mean 20.291
Statistical Analysis 2: Comparison: Fazirsiran 100 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -109.56, 95% CI 2-sided [-154.81 to -64.32], Standard Error of Mean 21.616
Statistical Analysis 3: Comparison: Fazirsiran 200 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -118.04, 95% CI 2-sided [-153.95 to -82.12], Standard Error of Mean 17.16

8. Secondary Outcome: Absolute Change From Baseline in Liver Z-AAT Insoluble Protein at Post-dose Biopsy for Participants With Fibrosis
Description: Post-dose biopsy includes all post-dose biopsy collected at Week 48 or Week 72 or Week 96.
Time Frame: Baseline, Week 48 (+/- 2 weeks), or Week 72 (+/- 4 weeks), or Week 96 (+/- 4 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nmol/g
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 8
nmol/g | -68.914 (80.725) | -150.145 (196.675) | -11.953 (18.602) | -7.038 (47.041)

9. Secondary Outcome: Percent Change From Baseline in Liver Z-AAT Insoluble Protein at Post-dose Biopsy for Participants With Fibrosis
Description: Post-dose biopsy includes all post-dose biopsy collected at Week 48 or Week 72 or Week 96.
Time Frame: Baseline, Week 48 (+/- 2 weeks), or Week 72 (+/- 4 weeks), or Week 96 (+/- 4 weeks)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 8
percentage change | -86.36 (60.305) | -72.44 (58.358) | -101.85 (47.495) | 91.35 (42.750)
Statistical Analysis 1: Comparison: Fazirsiran 25 mg vs Placebo; Test type: Superiority; p = 0.0247, ANCOVA — Model based summary statistics are from an analysis of covariance (ANCOVA) model with fixed effect factors treatment group and baseline insoluble liver Z-AAT protein as a covariate; LS Mean Difference = -180.7, 95% CI 2-sided [-335.77 to -25.64], Standard Error of Mean 74.087
Statistical Analysis 2: Comparison: Fazirsiran 100 mg vs Placebo; Test type: Superiority; p = 0.0382, ANCOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -163.79, 95% CI 2-sided [-317.65 to -9.93], Standard Error of Mean 73.513
Statistical Analysis 3: Comparison: Fazirsiran 200 mg vs Placebo; Test type: Superiority; p = 0.0064, ANCOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -193.2, 95% CI 2-sided [-325.25 to -61.15], Standard Error of Mean 63.089

10. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Alanine Aminotransferase (ALT) at Week 16 and Over Time Through End of Study (EOS)
Description: PDLB=post-dose liver biopsy
Time Frame: Baseline, Week 16, Week 16 + 24 hours (H), Weeks 28, 40, 48, 52, 64, 72, 76, 88, 96, 100, 112, 124, 136, 148, 160, Early Termination (up to 196 weeks), EOS (up to 208 weeks)
Population: Safety Analysis Set: all participants who received at least one dose of study drug; participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
U/L
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | -3.0 (9.17) | -2.4 (5.42) | -8.4 (15.88) | 1.7 (6.60)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -7.3 (11.93) | -3.8 (3.59) | -2.2 (2.86) | 0.8 (5.31)
  Week 28: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 28 | -10.7 (4.57) | -5.8 (9.56) | 0.6 (6.48) | 1.0 (6.91)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -4.6 (9.07) | -5.0 (8.78) | 3.1 (9.79) | -0.1 (4.66)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -10.5 (10.47) | 0.0 (16.00) | -2.2 (5.31) | 3.3 (7.71)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | -1.5 (12.31) | -6.0 (7.39) | 12.3 (33.80) | -0.4 (4.44)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -9.8 (8.50) | -14.3 (8.88) | -0.3 (8.30) | 5.7 (15.48)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -6.0 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -7.3 (3.06) | -14.8 (9.07) | 3.5 (8.24) | 7.7 (8.85)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -9.0 (3.46) | -18.5 (9.19) | 4.8 (4.97) | 6.2 (7.76)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -21.0 (5.66) | 12.0 (NA) — 1 participant analyzed | 10.0 (12.73)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -9.0 (2.83) | -21.5 (9.19) | 7.5 (7.78) | 1.3 (9.43)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -8.0 (NA) — 1 participant analyzed | -18.0 (7.07) | 8.0 (4.24) | -0.3 (6.43)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -18.0 (4.24) | 7.0 (NA) — 1 participant analyzed | 5.0 (11.53)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 4.0 (NA) — 1 participant analyzed | 8.3 (17.90)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 14
  Week 148 |  |  | 11.0 (NA) — 1 participant analyzed | 4.3 (14.98)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 23.0 (4.24)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -2.0 (9.90) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 7.0 (16.64) | -1.0 (5.66) | -0.5 (4.95) | -0.2 (5.45)

11. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: ALT at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | -9.6 (20.1) | -4.3 (19.9) | -15.3 (16.2) | 5.8 (16.1)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -15.7 (24.8) | -9.7 (8.9) | -10.8 (17.6) | 0.5 (13.3)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -27.4 (8.5) | -12.4 (25.1) | 2.0 (29.3) | 6.4 (21.9)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -11.2 (21.4) | -13.0 (24.0) | 4.0 (20.0) | 2.9 (18.3)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -21.7 (19.1) | -1.2 (38.2) | -4.8 (20.5) | 5.9 (15.2)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | -1.6 (32.9) | -15.2 (18.1) | 14.5 (28.5) | -1.4 (14.8)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -22.3 (20.3) | -33.3 (15.5) | 4.4 (35.8) | 11.0 (29.3)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -14.3 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -20.0 (7.0) | -33.7 (16.2) | 24.6 (43.6) | 26.3 (34.1)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -24.1 (0.0) | -39.8 (15.9) | 28.2 (32.6) | 20.7 (28.6)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -45.7 (7.5) | 60.0 (NA) — 1 participant analyzed | 44.8 (58.7)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -31.0 (9.8) | -46.4 (15.2) | 38.1 (38.1) | 9.9 (24.1)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -27.6 (NA) — 1 participant analyzed | -38.9 (11.3) | 41.4 (19.2) | 3.3 (24.7)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -39.3 (5.1) | 35.0 (NA) — 1 participant analyzed | 25.2 (49.4)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 20.0 (NA) — 1 participant analyzed | 40.1 (79.4)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 55.0 (NA) — 1 participant analyzed | 25.5 (61.4)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 88.8 (3.0)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -10.3 (65.0) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | 14.1 (38.7) | -6.8 (34.6) | -8.4 (15.0) | 4.7 (23.3)

12. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Aspartate Aminotransferase (AST) at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
U/L
  Week 16: number analyzed (Participants) | 9 | 7 | 8 | 13
  Week 16 | -2.9 (8.27) | -0.1 (4.02) | 1.1 (6.10) | 0.7 (5.23)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -7.7 (11.59) | 0.0 (2.58) | 0.3 (3.93) | -0.4 (3.81)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -7.4 (7.31) | -1.3 (4.68) | 10.2 (27.92) | 0.1 (5.49)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -2.9 (10.78) | 2.0 (17.55) | 2.9 (8.25) | -0.9 (3.65)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -12.0 (10.42) | 1.7 (4.16) | -1.0 (5.22) | 1.2 (6.40)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | -2.1 (9.89) | -0.9 (8.46) | 6.3 (15.92) | -0.9 (2.93)
  Week 64 | -8.8 (10.24) | -10.3 (10.40) | -0.7 (4.42) | 1.9 (7.70)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -3.0 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -6.3 (4.73) | -10.3 (8.85) | 3.2 (5.78) | 7.5 (7.20)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -6.7 (5.69) | -16.5 (12.02) | 3.8 (8.29) | 4.2 (6.57)
  PDLB at Week 96: number analyzed (Participants) | 0 | 1 | 1 | 2
  PDLB at Week 96 |  | -11.0 (NA) — 1 participant analyzed | 2.0 (NA) — 1 participant analyzed | 5.0 (5.66)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -7.5 (2.12) | -21.5 (13.44) | 1.5 (2.12) | 0.0 (4.76)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -10.0 (NA) — 1 participant analyzed | -19.0 (14.14) | 0.5 (0.71) | -2.0 (7.00)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -16.5 (10.61) | -1.0 (NA) — 1 participant analyzed | 2.7 (9.29)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | -2.0 (NA) — 1 participant analyzed | 6.7 (10.60)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 2.0 (NA) — 1 participant analyzed | 1.0 (11.14)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 10.5 (0.71)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -1.5 (4.95) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 4.7 (8.33) | 1.5 (6.36) | 1.5 (9.19) | -0.2 (3.96)

13. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: AST at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 16: number analyzed (Participants) | 9 | 7 | 8 | 13
  Week 16 | -8.3 (20.0) | 2.6 (16.4) | 3.5 (22.5) | 2.5 (14.3)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -16.9 (24.2) | 0.4 (7.8) | 1.5 (17.6) | 0.1 (9.8)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -19.3 (19.3) | -0.9 (14.5) | 26.8 (68.8) | 3.2 (17.4)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -4.7 (26.9) | 10.6 (43.4) | 8.3 (21.7) | -1.0 (11.4)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -27.1 (20.1) | 6.0 (12.5) | -2.0 (16.2) | 3.4 (19.2)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | -4.1 (27.2) | 1.9 (20.9) | 17.3 (40.3) | -2.8 (9.7)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -20.5 (23.3) | -21.4 (15.4) | -2.6 (16.8) | 9.5 (21.6)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -5.9 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -17.1 (12.7) | -22.2 (13.9) | 11.9 (22.6) | 30.3 (32.8)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -16.4 (10.1) | -30.6 (15.7) | 18.1 (34.7) | 21.1 (29.6)
  PDLB at Week 96: number analyzed (Participants) | 0 | 1 | 1 | 2
  PDLB at Week 96 |  | -26.8 (NA) — 1 participant analyzed | 7.4 (NA) — 1 participant analyzed | 31.9 (39.8)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -24.6 (9.1) | -40.5 (15.8) | 5.6 (7.9) | 5.2 (16.3)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -34.5 (NA) — 1 participant analyzed | -35.1 (18.7) | 2.5 (3.5) | 2.8 (27.0)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -31.0 (12.8) | -3.7 (NA) — 1 participant analyzed | 25.6 (53.1)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | -7.4 (NA) — 1 participant analyzed | 39.6 (70.4)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 7.4 (NA) — 1 participant analyzed | 21.8 (56.6)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 55.2 (25.7)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -7.3 (26.9) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 13.7 (24.6) | 10.5 (35.1) | -2.7 (31.5) | 0.7 (17.1)

14. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Alkaline Phosphatase (ALP) at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
U/L
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | -2.8 (9.98) | -4.3 (6.50) | -13.8 (14.26) | 4.9 (13.02)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -9.7 (8.62) | -1.0 (2.16) | -11.7 (14.83) | 3.6 (6.62)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | 0.6 (12.29) | -4.9 (6.88) | -8.4 (13.53) | 0.7 (5.51)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -1.1 (15.51) | -7.1 (6.36) | -8.3 (11.38) | 1.6 (7.43)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -10.5 (16.62) | -0.3 (1.15) | -2.8 (15.69) | 1.2 (2.56)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 52 | -3.0 (15.38) | -7.6 (8.26) | -3.9 (9.36) | 1.9 (6.01)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -8.3 (22.23) | -6.5 (8.96) | 0.4 (15.66) | 2.1 (9.25)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | 5.0 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -14.0 (23.39) | -9.0 (11.58) | 0.5 (11.50) | 6.5 (11.33)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -14.7 (21.13) | -16.5 (23.33) | 3.0 (21.25) | 8.4 (8.02)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -11.5 (13.44) | 2.0 (NA) — 1 participant analyzed | 7.0 (19.80)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -23.0 (26.87) | -11.5 (17.68) | -2.0 (2.83) | 8.8 (12.04)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -4.0 (NA) — 1 participant analyzed | -6.0 (11.31) | -2.0 (4.24) | 5.0 (13.75)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -4.0 (5.66) | 4.0 (NA) — 1 participant analyzed | 4.3 (9.24)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 2.0 (NA) — 1 participant analyzed | 7.0 (25.16)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 15.0 (NA) — 1 participant analyzed | 11.0 (26.46)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 23.0 (26.87)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -0.5 (17.68) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | 1.8 (10.40) | -6.0 (0.00) | 5.0 (9.90) | 3.4 (11.76)

15. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: ALP at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | -0.5 (12.8) | -5.6 (8.7) | -17.7 (16.0) | 5.8 (14.7)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -8.9 (6.1) | -1.2 (2.8) | -14.8 (16.8) | 5.9 (10.0)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | 5.5 (20.1) | -6.4 (9.3) | -10.5 (16.1) | 1.0 (7.2)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | 2.0 (16.9) | -9.3 (8.2) | -10.4 (14.9) | 2.2 (10.4)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -8.5 (13.9) | -0.4 (1.5) | -3.3 (23.5) | 1.7 (3.7)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 52 | 0.1 (17.0) | -9.7 (11.7) | -4.9 (13.5) | 2.7 (8.3)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -5.6 (18.4) | -8.3 (10.8) | -0.2 (22.5) | 3.9 (11.0)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | 7.1 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -11.2 (18.2) | -11.4 (13.5) | 0.7 (18.1) | 8.0 (13.3)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -12.5 (15.9) | -19.6 (27.8) | 3.2 (30.3) | 10.6 (9.5)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -13.9 (15.7) | 2.9 (NA) — 1 participant analyzed | 7.6 (22.6)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -19.4 (19.4) | -13.6 (21.2) | -2.5 (3.6) | 10.1 (13.4)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -5.6 (NA) — 1 participant analyzed | -6.9 (13.8) | -2.4 (5.5) | 5.7 (15.6)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -4.8 (6.7) | 5.8 (NA) — 1 participant analyzed | 4.7 (10.5)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 2.9 (NA) — 1 participant analyzed | 6.8 (29.3)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 21.7 (NA) — 1 participant analyzed | 11.5 (30.8)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 26.0 (30.0)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 4.6 (26.1) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | 7.8 (18.2) | -7.2 (1.8) | 7.1 (13.9) | 5.3 (12.3)

16. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Gamma Glutamyl Transferase (GGT) at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: Baseline, Week 16, Week 16 + 24 hours (H), Weeks 28, 40, 48, 52, 64, 72, 76, 88, 96, 100, 112, 124,136, 148, 160, Early Termination (up to 196 weeks), EOS (up to 208 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
U/L
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | 2.8 (11.48) | -4.3 (5.90) | -9.1 (16.06) | 7.0 (14.88)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | -3.7 (16.80) | -4.8 (4.35) | -4.3 (4.93) | 1.1 (4.62)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -3.5 (11.99) | -5.3 (5.57) | -4.1 (9.65) | 0.6 (8.47)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | 5.3 (31.24) | -3.8 (9.29) | 0.9 (16.88) | 0.6 (7.69)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -13.5 (23.67) | -5.3 (4.16) | -5.3 (10.17) | -0.5 (10.48)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | 7.3 (36.39) | -4.3 (11.13) | 6.8 (27.79) | 1.7 (6.64)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -16.0 (13.22) | -13.0 (14.14) | 2.7 (19.04) | 9.3 (22.13)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -3.0 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -20.3 (28.36) | -13.3 (15.48) | -3.3 (11.04) | -0.3 (10.19)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -17.0 (29.51) | -19.0 (25.46) | 2.0 (7.81) | 7.2 (4.97)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -25.5 (14.85) | 5.0 (NA) — 1 participant analyzed | 3.5 (0.71)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -25.0 (28.28) | -24.5 (21.92) | 6.5 (4.95) | -2.3 (14.29)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | 0.0 (NA) — 1 participant analyzed | -21.5 (9.19) | 5.5 (4.95) | 4.3 (10.41)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -50.4 (2.6) | 8.0 (NA) — 1 participant analyzed | 1.7 (9.61)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 7.0 (NA) — 1 participant analyzed | 5.0 (7.55)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 10.0 (NA) — 1 participant analyzed | -0.3 (11.59)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 3.0 (4.24)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 5.0 (4.24) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | 22.5 (45.68) | -0.5 (0.71) | -19.5 (27.58) | 0.6 (5.59)

17. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: GGT at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | 5.9 (18.9) | -9.7 (12.7) | -14.8 (18.5) | 13.9 (31.0)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | 0.8 (32.2) | -9.1 (8.6) | -13.2 (13.6) | 4.7 (15.4)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -2.2 (21.5) | -12.0 (11.7) | -3.2 (22.2) | 6.8 (21.5)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | 14.4 (52.4) | -6.4 (18.3) | -1.7 (31.6) | 7.4 (14.4)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -8.9 (36.3) | -13.3 (7.2) | -10.4 (30.9) | 8.1 (17.6)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | 26.7 (69.5) | -3.5 (25.1) | 6.2 (35.2) | 5.1 (15.3)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -23.0 (6.7) | -22.8 (17.8) | 20.7 (69.3) | 13.1 (24.9)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -6.7 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -22.2 (13.6) | -23.1 (18.9) | -0.9 (38.4) | 9.5 (13.3)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | 13.7 (21.1) | -26.8 (34.7) | 15.6 (39.5) | 17.9 (15.1)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -42.0 (11.2) | 25.0 (NA) — 1 participant analyzed | 11.9 (2.7)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -23.4 (11.7) | -38.0 (24.8) | 33.8 (22.9) | 6.1 (24.2)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | 0.0 (NA) — 1 participant analyzed | -36.5 (3.4) | 28.4 (23.5) | 16.0 (32.9)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -50.4 (2.6) | 40.0 (NA) — 1 participant analyzed | 8.1 (28.7)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 35.0 (NA) — 1 participant analyzed | 18.0 (23.4)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 50.0 (NA) — 1 participant analyzed | 2.9 (33.3)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 10.0 (14.1)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 30.7 (32.1) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | 39.2 (78.5) | -2.2 (3.1) | -17.1 (24.2) | 6.7 (18.8)

18. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Total Bilirubin at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
mg/dL
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | 0.079 (0.146) | 0.098 (0.369) | -0.051 (0.241) | -0.004 (0.208)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | 0.060 (0.075) | 0.163 (0.456) | -0.040 (0.182) | -0.118 (0.105)
  Week 28: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 28 | 0.109 (0.149) | 0.171 (0.470) | 0.053 (0.230) | 0.012 (0.272)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | 0.083 (0.115) | 0.164 (0.437) | 0.017 (0.092) | 0.062 (0.434)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | 0.043 (0.109) | -0.070 (0.594) | 0.098 (0.252) | -0.085 (0.178)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 52 | -0.023 (0.203) | 0.129 (0.362) | 0.086 (0.165) | 0.099 (0.230)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | 0.020 (0.210) | 0.188 (0.235) | 0.006 (0.208) | -0.086 (0.188)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -0.420 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | 0.110 (0.105) | 0.248 (0.357) | -0.043 (0.206) | -0.018 (0.198)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | 0.247 (0.375) | 0.105 (0.035) | 0.002 (0.131) | -0.050 (0.131)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | 0.020 (0.127) | 0.170 (NA) — 1 participant analyzed | 0.065 (0.035)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -0.040 (0.099) | -0.055 (0.106) | 0.090 (0.042) | 0.003 (0.203)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -0.020 (NA) — 1 participant analyzed | -0.010 (0.269) | 0.100 (0.141) | -0.060 (0.249)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -0.190 (0.071) | 0.130 (NA) — 1 participant analyzed | -0.037 (0.085)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 0.100 (NA) — 1 participant analyzed | 0.003 (0.185)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 0.070 (NA) — 1 participant analyzed | -0.087 (0.199)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | -0.090 (0.028)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -0.010 (0.014) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 0.170 (0.123) | 0.050 (0.113) | 0.025 (0.205) | 0.154 (0.082)

19. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: Total Bilirubin at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 16: number analyzed (Participants) | 9 | 8 | 8 | 14
  Week 16 | 19.2 (38.5) | 15.6 (41.7) | 3.4 (44.1) | 1.0 (28.0)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 9
  Week 16 + 24 H | 16.4 (19.2) | 25.3 (49.7) | 3.1 (33.1) | -16.3 (12.6)
  Week 28: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 28 | 26.7 (36.1) | 27.8 (51.4) | 15.8 (36.8) | 1.3 (37.5)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | 20.6 (27.8) | 30.2 (51.4) | 10.0 (21.6) | 7.8 (46.4)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | 11.8 (27.8) | 10.8 (68.2) | 36.5 (52.2) | -10.9 (29.4)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 13
  Week 52 | -8.3 (36.6) | 27.5 (48.8) | 25.4 (29.4) | 15.5 (36.4)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | 10.3 (51.0) | 28.5 (38.0) | 10.0 (35.7) | -13.3 (28.1)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -60.0 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | 18.1 (16.1) | 40.1 (57.1) | 0.3 (31.6) | -1.0 (33.2)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | 38.0 (53.7) | 13.1 (1.7) | 5.4 (29.3) | -7.6 (21.4)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | 0.8 (15.9) | 39.5 (NA) — 1 participant analyzed | 9.2 (1.7)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -11.9 (25.2) | -8.6 (15.3) | 25.1 (4.0) | 0.4 (31.6)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -5.4 (NA) — 1 participant analyzed | -5.0 (35.1) | 37.0 (52.4) | -5.8 (30.8)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -23.6 (3.9) | 30.2 (NA) — 1 participant analyzed | -5.7 (12.4)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 23.3 (NA) — 1 participant analyzed | 4.4 (25.2)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 16.3 (NA) — 1 participant analyzed | -7.6 (29.7)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | -13.4 (0.9)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -2.9 (4.2) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 41.8 (36.4) | 11.5 (26.4) | 25.0 (69.2) | 26.8 (16.6)

20. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Direct Bilirubin at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
mg/dL
  Week 16: number analyzed (Participants) | 8 | 7 | 7 | 12
  Week 16 | 0.016 (0.049) | -0.006 (0.095) | 0.005 (0.094) | 0.010 (0.061)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 8
  Week 16 + 24 H | 0.013 (0.029) | 0.055 (0.157) | -0.030 (0.081) | -0.028 (0.041)
  Week 28: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 28 | 0.029 (0.055) | 0.039 (0.140) | 0.004 (0.062) | 0.008 (0.073)
  Week 40: number analyzed (Participants) | 7 | 8 | 9 | 13
  Week 40 | 0.026 (0.050) | 0.045 (0.160) | -0.005 (0.063) | 0.020 (0.125)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 5
  PDLB at Week 48 | -0.005 (0.041) | -0.080 (0.210) | 0.007 (0.087) | -0.038 (0.065)
  Week 52: number analyzed (Participants) | 7 | 8 | 9 | 13
  Week 52 | -0.024 (0.080) | 0.034 (0.107) | 0.015 (0.052) | 0.031 (0.058)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -0.008 (0.081) | 0.053 (0.061) | -0.007 (0.076) | -0.019 (0.043)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -46.2 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | 0.027 (0.029) | 0.098 (0.069) | -0.033 (0.073) | 0.027 (0.057)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | 0.053 (0.114) | 0.070 (0.014) | -0.007 (0.043) | 0.012 (0.026)
  PDLB at Week 96: number analyzed (Participants) | 0 | 1 | 1 | 2
  PDLB at Week 96 |  | 0.030 (NA) — 1 participant analyzed | 0.080 (NA) — 1 participant analyzed | 0.045 (0.035)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | 0.000 (0.028) | 0.010 (0.014) | 0.050 (0.028) | 0.018 (0.052)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | 0.020 (NA) — 1 participant analyzed | 0.025 (0.049) | 0.055 (0.035) | 0.007 (0.061)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -0.040 (0.057) | 0.070 (NA) — 1 participant analyzed | 0.020 (0.035)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 0.030 (NA) — 1 participant analyzed | 0.013 (0.046)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 0.050 (NA) — 1 participant analyzed | -0.003 (0.090)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 0.015 (0.007)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 0.005 (0.007) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 0.050 (0.060) | 0.010 (0.028) | 0.028 (0.138) | 0.053 (0.044)

21. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: Direct Bilirubin at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
percentage change
  Week 16: number analyzed (Participants) | 8 | 7 | 7 | 12
  Week 16 | 5.9 (30.1) | 1.5 (31.2) | 29.1 (67.6) | 15.1 (58.9)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 6 | 8
  Week 16 + 24 H | 11.0 (16.4) | 22.4 (50.9) | -0.1 (33.0) | -8.8 (17.0)
  Week 28: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 28 | 19.0 (28.3) | 15.4 (37.3) | 21.2 (61.9) | 10.1 (44.6)
  Week 40: number analyzed (Participants) | 7 | 8 | 9 | 13
  Week 40 | 17.9 (27.5) | 16.7 (44.9) | 15.5 (47.6) | 14.3 (50.2)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 5
  PDLB at Week 48 | 2.9 (19.5) | -9.9 (63.0) | 19.3 (48.7) | -11.9 (23.9)
  Week 52: number analyzed (Participants) | 7 | 8 | 9 | 13
  Week 52 | -12.1 (34.3) | 17.8 (35.1) | 25.1 (47.0) | 19.6 (38.5)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | 4.4 (39.7) | 18.9 (26.7) | 8.2 (37.3) | -8.6 (16.7)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -46.2 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | 9.9 (7.4) | 33.4 (20.2) | -5.4 (30.0) | 11.4 (21.5)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | 18.2 (35.0) | 24.9 (14.0) | -3.3 (30.3) | 5.6 (12.1)
  PDLB at Week 96: number analyzed (Participants) | 0 | 1 | 1 | 2
  PDLB at Week 96 |  | 7.5 (NA) — 1 participant analyzed | 53.3 (NA) — 1 participant analyzed | 17.1 (10.0)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -3.8 (16.3) | 4.3 (6.1) | 37.0 (13.7) | 7.5 (23.2)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | 15.4 (NA) — 1 participant analyzed | 5.3 (13.7) | 46.4 (37.3) | 4.1 (22.5)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -10.0 (14.1) | 46.7 (NA) — 1 participant analyzed | 7.7 (13.3)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 20.0 (NA) — 1 participant analyzed | 7.2 (18.3)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 33.3 (NA) — 1 participant analyzed | 3.4 (38.5)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 6.7 (4.6)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 2.4 (3.4) |
  End of Study: number analyzed (Participants) | 3 | 2 | 2 | 5
  End of Study | 34.3 (45.6) | 5.4 (14.7) | 96.1 (185.5) | 40.8 (46.7)

22. Secondary Outcome: Absolute Change From Baseline in Liver Function Tests: Prothrombin International Normalized Ratio at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
ratio
  Week 16 | -0.012 (0.054) | -0.006 (0.093) | 0.011 (0.068) | 0.055 (0.180)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 7 | 9
  Week 16 + 24 H | 0.047 (0.111) | -0.085 (0.093) | -0.017 (0.117) | 0.036 (0.104)
  Week 28: number analyzed (Participants) | 8 | 8 | 8 | 14
  Week 28 | -0.054 (0.148) | -0.059 (0.109) | -0.040 (0.107) | -0.014 (0.167)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -0.021 (0.113) | -0.024 (0.099) | -0.022 (0.125) | 0.034 (0.143)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -0.038 (0.054) | -0.067 (0.150) | -0.023 (0.121) | 0.022 (0.048)
  Week 52: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 52 | -0.094 (0.139) | -0.053 (0.057) | -0.034 (0.076) | -0.002 (0.076)
  Week 64: number analyzed (Participants) | 4 | 3 | 7 | 9
  Week 64 | -0.038 (0.089) | -0.100 (0.082) | -0.043 (0.130) | 0.012 (0.055)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | 0.040 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -0.033 (0.049) | -0.110 (0.130) | -0.065 (0.136) | 0.020 (0.046)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -0.053 (0.040) | -0.225 (0.177) | -0.004 (0.083) | 0.038 (0.026)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -0.195 (0.134) | 0.090 (NA) — 1 participant analyzed | 0.045 (0.078)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | 0.000 (0.014) | -0.225 (0.163) | -0.020 (0.099) | 0.063 (0.045)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | 0.050 (NA) — 1 participant analyzed | -0.240 (0.184) | 0.035 (0.078) | 0.047 (0.083)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -0.175 (0.247) | 0.050 (NA) — 1 participant analyzed | 0.053 (0.021)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 0.070 (NA) — 1 participant analyzed | 0.043 (0.032)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 0.080 (NA) — 1 participant analyzed | 0.040 (0.026)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 0.070 (0.042)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 0.045 (0.092) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | -0.115 (0.170) | -0.045 (0.049) | -0.035 (0.021) | -0.106 (0.149)

23. Secondary Outcome: Percent Change From Baseline in Liver Function Tests: Prothrombin International Normalized Ratio at Week 16 and Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 16 | -1.0 (4.8) | -0.7 (7.7) | 1.2 (6.4) | 2.6 (8.6)
  Week 16 + 24 H: number analyzed (Participants) | 3 | 4 | 7 | 9
  Week 16 + 24 H | 4.4 (10.3) | -7.0 (6.9) | -1.0 (10.2) | 3.5 (9.9)
  Week 28: number analyzed (Participants) | 8 | 8 | 8 | 14
  Week 28 | -3.9 (11.8) | -4.9 (8.5) | -3.3 (9.1) | 1.2 (8.7)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -1.2 (9.6) | -1.6 (7.8) | -1.6 (11.3) | 3.7 (13.0)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -3.2 (4.7) | -5.5 (13.3) | -1.5 (10.3) | 2.2 (4.8)
  Week 52: number analyzed (Participants) | 7 | 8 | 9 | 14
  Week 52 | -7.7 (10.2) | -4.7 (4.9) | -2.9 (6.3) | 0.3 (6.9)
  Week 64: number analyzed (Participants) | 4 | 3 | 7 | 9
  Week 64 | -3.2 (7.9) | -8.4 (7.1) | -3.2 (11.4) | 1.3 (5.3)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | 3.9 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -2.8 (4.0) | -8.8 (9.9) | -5.3 (11.8) | 2.0 (4.6)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -4.7 (3.1) | -17.9 (12.5) | -0.3 (8.0) | 3.7 (2.4)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -15.6 (9.2) | 9.0 (NA) — 1 participant analyzed | 4.6 (7.8)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | 0.0 (1.4) | -18.0 (11.3) | -1.8 (9.6) | 6.2 (4.5)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | 4.9 (NA) — 1 participant analyzed | -19.1 (12.9) | 3.5 (7.7) | 4.7 (8.4)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -13.4 (18.9) | 5.0 (NA) — 1 participant analyzed | 5.3 (2.1)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | 7.0 (NA) — 1 participant analyzed | 4.3 (3.3)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | 8.0 (NA) — 1 participant analyzed | 3.9 (2.5)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 7.0 (4.3)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | 4.8 (9.4) |
  End of Study: number analyzed (Participants) | 4 | 2 | 2 | 5
  End of Study | -9.1 (12.7) | -4.3 (4.9) | -3.6 (2.0) | -5.8 (4.7)

24. Secondary Outcome: Absolute Change in Serum Z-AAT Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: Baseline, Weeks 2, 4, 6, 16, 28, 40, 48, 52, 64, 72, 76, 88, 96, 100, 112, 124, 136, 148, 160, Early Termination (up to 196 weeks), EOS (up to 208 weeks)
Population: Full Analysis Set: All randomized participants who received at least one dose of study drug; participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
μg/mL
  Week 2: number analyzed (Participants) | 9 | 7 | 9 | 14
  Week 2 | -125.511 (59.955) | -156.714 (58.127) | -169.044 (40.328) | 16.929 (37.723)
  Week 4 | -146.267 (68.511) | -178.413 (58.821) | -181.389 (41.857) | -0.429 (18.826)
  Week 6 | -176.100 (47.242) | -192.719 (65.087) | -188.781 (43.539) | 7.000 (26.712)
  Week 16: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 16 | -158.650 (50.266) | -185.213 (58.059) | -182.240 (45.710) | 10.286 (29.374)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -123.288 (62.112) | -174.275 (57.293) | -175.136 (52.838) | -0.500 (25.035)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -122.288 (70.057) | -165.763 (59.312) | -164.629 (63.830) | 1.429 (20.137)
  PDLB at Week 48 | -189.850 (64.556) | -150.900 (17.521) | -194.535 (51.128) | 14.333 (38.754)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 52 | -116.188 (72.983) | -157.300 (56.023) | -165.741 (64.535) | -13.643 (36.527)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -187.325 (94.397) | -191.150 (80.589) | -190.284 (45.070) | 0.333 (27.208)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -6.00 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -164.067 (65.875) | -189.225 (91.259) | -177.060 (49.718) | -9.500 (20.907)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -142.767 (89.632) | -260.200 (82.166) | -186.116 (44.539) | -1.800 (28.490)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -271.100 (90.793) | -194.160 (NA) — 1 participant analyzed | -35.000 (15.556)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -204.650 (18.597) | -244.100 (91.358) | -187.650 (3.323) | -60.725 (84.824)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -233.000 (NA) — 1 participant analyzed | -263.100 (91.358) | -182.550 (3.182) | -22.333 (22.679)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -237.650 (102.743) | -183.000 (NA) — 1 participant analyzed | -26.000 (22.271)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | -183.300 (NA) — 1 participant analyzed | -8.000 (22.650)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | -89.1 (NA) — 1 participant analyzed | 9.333 (11.719)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 7.500 (9.192)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -192.240 (81.657) |
  End of Study: number analyzed (Participants) | 4 | 3 | 2 | 4
  End of Study | -42.750 (7.089) | -103.533 (3.443) | -39.000 (1.414) | 19.750 (30.966)

25. Secondary Outcome: Percent Change in Serum Z-AAT Over Time Through EOS
Description: PDLB=post-dose liver biopsy
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 14
percentage change
  Week 2: number analyzed (Participants) | 9 | 7 | 9 | 14
  Week 2 | -50.8 (21.9) | -69.9 (11.4) | -85.5 (4.8) | 10.0 (23.8)
  Week 4 | -60.0 (24.6) | -82.2 (7.1) | -91.8 (2.5) | 0.5 (8.7)
  Week 6 | -71.9 (14.0) | -88.4 (5.0) | -95.5 (1.9) | 3.4 (11.4)
  Week 16: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 16 | -62.4 (17.0) | -85.7 (7.6) | -91.9 (5.8) | 4.3 (12.2)
  Week 28: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 28 | -48.2 (20.6) | -80.6 (7.9) | -87.6 (10.4) | 0.1 (11.2)
  Week 40: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 40 | -48.3 (23.4) | -76.5 (10.5) | -81.3 (18.8) | 0.3 (9.2)
  PDLB at Week 48: number analyzed (Participants) | 4 | 3 | 6 | 6
  PDLB at Week 48 | -73.9 (16.7) | -89.2 (2.5) | -93.9 (5.0) | 8.7 (19.0)
  Week 52: number analyzed (Participants) | 8 | 8 | 9 | 14
  Week 52 | -45.9 (24.7) | -73.0 (12.9) | -82.1 (20.5) | -5.3 (14.9)
  Week 64: number analyzed (Participants) | 4 | 4 | 7 | 9
  Week 64 | -70.1 (23.5) | -77.6 (9.5) | -92.2 (5.7) | 2.1 (12.3)
  PDLB at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 1
  PDLB at Week 72 |  |  |  | -2.4 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 3 | 4 | 6 | 6
  Week 76 | -71.8 (19.6) | -75.1 (9.0) | -88.8 (10.1) | -2.4 (9.3)
  Week 88: number analyzed (Participants) | 3 | 2 | 5 | 5
  Week 88 | -60.1 (32.6) | -77.8 (7.2) | -90.3 (6.3) | 0.5 (11.4)
  PDLB at Week 96: number analyzed (Participants) | 0 | 2 | 1 | 2
  PDLB at Week 96 |  | -80.9 (9.1) | -95.6 (NA) — 1 participant analyzed | -11.7 (4.2)
  Week 100: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 100 | -82.5 (10.1) | -72.5 (11.2) | -93.8 (0.3) | -21.3 (29.6)
  Week 112: number analyzed (Participants) | 1 | 2 | 2 | 3
  Week 112 | -91.7 (NA) — 1 participant analyzed | -78.4 (9.9) | -91.3 (3.5) | -8.4 (9.2)
  Week 124: number analyzed (Participants) | 0 | 2 | 1 | 3
  Week 124 |  | -70.1 (15.2) | -90.1 (NA) — 1 participant analyzed | -9.9 (9.1)
  Week 136: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 136 |  |  | -90.3 (NA) — 1 participant analyzed | -3.2 (8.8)
  Week 148: number analyzed (Participants) | 0 | 0 | 1 | 3
  Week 148 |  |  | -89.1 (NA) — 1 participant analyzed | 3.1 (4.1)
  Week 160: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 160 |  |  |  | 2.4 (2.9)
  Early Termination: number analyzed (Participants) | 0 | 0 | 2 | 0
  Early Termination |  |  | -91.7 (8.5) |
  End of Study: number analyzed (Participants) | 4 | 3 | 2 | 4
  End of Study | -18.0 (2.7) | -53.8 (6.6) | -23.4 (0.1) | 9.1 (12.4)

26. Secondary Outcome: Pharmacokinetics (PK): ARO-AAT Plasma Concentration Summary for the Double-Blind Phase
Time Frame: Fazirsiran participants without fibrosis: Pre-dose, 1 hour, 2 hour, 24 hours post-dose on Day 1 (+/- 1 day). Fazirsiran participants with fibrosis: Pre-dose, 1 hour, 2 hours, 24 hours post-dose on Day 1 and Week 16 (+/- 1 day).
Population: PK Population: all Full Analysis Set participants who have at least 1 measurable plasma concentration data; participants with an assessment at given time point. Data not collected Week 16 for participants with no fibrosis per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Fazirsiran 25 mg: Participants With No Fibrosis: Participants with no fibrosis: Fazirsiran 25 mg administered on Day 1 and Week 4.
- Fazirsiran 25 mg: Participants With Fibrosis: Participants with fibrosis: Fazirsiran 25 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
- Fazirsiran 100 mg: Participants With No Fibrosis: Participants with no fibrosis: Fazirsiran 100 mg administered on Day 1 and Week 4.
- Fazirsiran 100 mg: Participants With Fibrosis: Participants with fibrosis: Fazirsiran 100 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
- Fazirsiran 200 mg: Participants With No Fibrosis: Participants with no fibrosis: Fazirsiran 200 mg administered on Day 1 and Week 4.
- Fazirsiran 200 mg: Participants With Fibrosis: Participants with fibrosis: Fazirsiran 200 mg administered on Day 1, Week 4, and Week 16, then every 12 weeks up to 18 total doses.
Arm/Group | Fazirsiran 25 mg: Participants With No Fibrosis | Fazirsiran 25 mg: Participants With Fibrosis | Fazirsiran 100 mg: Participants With No Fibrosis | Fazirsiran 100 mg: Participants With Fibrosis | Fazirsiran 200 mg: Participants With No Fibrosis | Fazirsiran 200 mg: Participants With Fibrosis
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 2 | 7
ng/mL
  Day 1, Pre-Dose | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 1, 1 hour (h) | 29.9 (75.6) | 50.6 (66.8) | 190.0 (17.9) | 173.0 (25.7) | 495.0 (71.8) | 356.0 (75.9)
  Day 1, 2h | 35.0 (83.0) | 60.7 (72.5) | 208.0 (11.6) | 199.0 (32.2) | 537.0 (81.9) | 471.0 (56.5)
  Day 1, 24h: number analyzed (Participants) | 4 | 4 | 3 | 5 | 2 | 6
  Day 1, 24h | 9.92 (99.6) | 6.33 (176.0) | 69.0 (88.4) | 26.6 (59.1) | 11.7 (17100) | 27.7 (612.0)
  Week 16, Pre-Dose: number analyzed (Participants) | 1 | 4 | 3 | 5 | 1 | 7
  Week 16, Pre-Dose | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 16, 1h: number analyzed (Participants) | 0 | 3 | 0 | 5 | 0 | 7
  Week 16, 1h |  | 38.1 (75.3) |  | 38.1 (75.3) |  | 396.0 (64.9)
  Week 16, 2h: number analyzed (Participants) | 0 | 3 | 0 | 5 | 0 | 7
  Week 16, 2h |  | 45.1 (70.1) |  | 45.1 (70.1) |  | 487.0 (62.5)
  Week 16, 24h: number analyzed (Participants) | 0 | 3 | 0 | 5 | 0 | 7
  Week 16, 24h |  | 3.64 (123.0) |  | 3.64 (123.0) |  | 104.0 (26.2)

27. Secondary Outcome: Number of Participants Positive for Anti-Drug Antibodies to Fazirsiran
Description: PDLB=post-dose liver biopsy
Time Frame: Baseline, Weeks 4, 16, 28, 40, 48, 52, 64, 76, 88, 96, 100, 112, 124, 136, 148 or Early Termination (up to 148 weeks)
Population: Safety Analysis Set: all participants who received at least one dose of fazirsiran; participants with an assessment at given time point
Measure: Count of Participants; unit: Participants
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg
Number analyzed (Participants) | 9 | 8 | 9
Participants
  Baseline | 0 | 2 | 2
  Week 4 | 0 | 1 | 2
  Week 16: number analyzed (Participants) | 7 | 8 | 9
  Week 16 | 0 | 1 | 2
  Week 28: number analyzed (Participants) | 7 | 8 | 8
  Week 28 | 0 | 2 | 1
  Week 40: number analyzed (Participants) | 8 | 8 | 9
  Week 40 | 0 | 2 | 2
  PDLB at Week 48: number analyzed (Participants) | 1 | 0 | 1
  PDLB at Week 48 | 0 |  | 0
  Week 52: number analyzed (Participants) | 6 | 5 | 7
  Week 52 | 0 | 1 | 0
  Week 64: number analyzed (Participants) | 4 | 4 | 7
  Week 64 | 0 | 0 | 0
  Week 76: number analyzed (Participants) | 3 | 4 | 6
  Week 76 | 0 | 1 | 0
  Week 88: number analyzed (Participants) | 3 | 2 | 5
  Week 88 | 0 | 0 | 0
  PDLB at Week 96: number analyzed (Participants) | 0 | 0 | 1
  PDLB at Week 96 |  |  | 0
  Week 100: number analyzed (Participants) | 2 | 2 | 2
  Week 100 | 0 | 0 | 0
  Week 112: number analyzed (Participants) | 1 | 2 | 2
  Week 112 | 0 | 0 | 1
  Week 124: number analyzed (Participants) | 0 | 2 | 1
  Week 124 |  | 0 | 1
  Week 136: number analyzed (Participants) | 0 | 0 | 9
  Week 136 |  |  | 1
  Week 148: number analyzed (Participants) | 0 | 0 | 1
  Week 148 |  |  | 1
  Early Termination: number analyzed (Participants) | 0 | 0 | 2
  Early Termination |  |  | 0

28. Secondary Outcome: Percentage of Participants With Shifts From Baseline in METAVIR Fibrosis Stage at Post-Dose Biopsy for Participants With Fibrosis
Description: The METAVIR scoring system is a system used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy. The stage represents the amount of fibrosis or scarring: 0= no fibrosis; 1=portal fibrosis without septa; 2=portal fibrosis with few septa; 3=numerous septa without cirrhosis; 4=cirrhosis. A higher score indicates a worse condition.
Time Frame: Baseline, Post-dose at Weeks 48 (+/- 2 weeks) or Week 72 (+/- 4 weeks) or Week 96 (+/- 4 weeks)
Population: Biopsy Analysis Set: All randomized participants who received at least one dose of study drug and had at least one central read histology biopsy result; participants eligible to meet the defined criteria. (For example, participants with baseline METAVIR fibrosis score 0 are not eligible for improvement; participants with baseline METAVIR fibrosis score 4 are not eligible for worsening.)
Measure: Number; unit: percentage of participants
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo
Number analyzed (Participants) | 4 | 5 | 7 | 9
percentage of participants
  >= 1-point improvement from baseline: number analyzed (Participants) | 3 | 5 | 6 | 8
  >= 1-point improvement from baseline | 66.7 | 40.0 | 50.0 | 37.5
  no change from baseline | 25.0 | 60.0 | 14.3 | 44.4
  >= 1-point worsening from baseline | 25.0 | 0.0 | 42.9 | 22.2

ADVERSE EVENTS:
Time Frame: Participants without fibrosis: for a maximum duration of follow up of 66 weeks. Participants with evidence of fibrosis: for a maximum duration of follow up of 210 weeks.
Arm/Group | Fazirsiran 25 mg | Fazirsiran 100 mg | Fazirsiran 200 mg | Placebo | Fazirsiran 25 mg DB/200 mg OL | Fazirsiran 100 mg DB/200 mg OL | Fazirsiran 200 mg DB/200 mg OL | Placebo DB / Fazirsiran 200 mg OL
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/14 | 0/4 | 0/5 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 2/9 | 3/14 | 1/4 | 1/5 | 1/5 | 1/9
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8 | 9/9 | 14/14 | 4/4 | 4/5 | 3/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fazirsiran 25 mg (N=9) | Fazirsiran 100 mg (N=8) | Fazirsiran 200 mg (N=9) | Placebo (N=14) | Fazirsiran 25 mg DB/200 mg OL (N=4) | Fazirsiran 100 mg DB/200 mg OL (N=5) | Fazirsiran 200 mg DB/200 mg OL (N=5) | Placebo DB / Fazirsiran 200 mg OL (N=9)
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fazirsiran 25 mg (N=9) | Fazirsiran 100 mg (N=8) | Fazirsiran 200 mg (N=9) | Placebo (N=14) | Fazirsiran 25 mg DB/200 mg OL (N=4) | Fazirsiran 100 mg DB/200 mg OL (N=5) | Fazirsiran 200 mg DB/200 mg OL (N=5) | Placebo DB / Fazirsiran 200 mg OL (N=9)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left atrial enlargement (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hamartoma (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic steatosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 7 | 2 | 0 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Atypical mycobacterial pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatophytosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incision site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pertussis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site induration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Forced vital capacity decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung diffusion test decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spirometry abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 2 | 4 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breathing-related sleep disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Withdrawal hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT03945292/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03945292/SAP_001.pdf